CLINICAL TRIAL: NCT06854289
Title: Comparison of the Impact of Physical Activity Attitude on Physical Activity Level and Postural Awareness Between Physiotherapy and Rehabilitation Department Students and Software Engineering Department Students
Brief Title: Comparison of the Impact of Physical Activity Attitude Between Different Department University Students
Status: Not yet recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Öznur TAŞAR, Physiotherapy and Rehabilitation, Firat University
Other Study IDs: 2024/15-33
Record Dates: First submitted 2025-02-23; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Physical Activity Level; Postural Awareness; Physical Activity Attitude; University Students
Keywords: Physical activity level; Postural Awareness; Physical Activity Attitude; University Students

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Physiotherapy and rehabilitation student
- Software engineering student

SUMMARY:
In recent years, the level of physical activity among university students has been steadily decreasing, and young people are leading a sedentary lifestyle. The aim of this study is to evaluate and compare the perspectives and attitudes towards physical activity of students from the Physiotherapy and Rehabilitation department, who are expected to have awareness of physical activity due to their undergraduate education, with students from the Software Engineering department, who do not receive education on this subject. The study will also investigate how these perspectives and attitudes affect their level of physical activity and postural awareness.Software Engineering students and Physiotherapy and Rehabilitation department students between the ages of 20-25, studying in the 3rd and 4th grades at Fırat University, will be included in the study. A questionnaire regarding the sociodemographic characteristics of the participants, Physical Activity Attitude Scale, International Physical Activity Survey Short Form, Postural Awareness Scale Turkish Version will be used as data collection tools.

DETAILED DESCRIPTION:
In recent years, the level of physical activity among university students has been steadily decreasing, and young people are leading a sedentary lifestyle. The aim of this study is to evaluate and compare the perspectives and attitudes towards physical activity of students from the Physiotherapy and Rehabilitation department, who are expected to have awareness of physical activity due to their undergraduate education, with students from the Software Engineering department, who do not receive education on this subject. The study will also investigate how these perspectives and attitudes affect their level of physical activity and postural awareness.Software Engineering students and Physiotherapy and Rehabilitation department students between the ages of 20-25, studying in the 3rd and 4th grades at Fırat University, will be included in the study. A questionnaire regarding the sociodemographic characteristics of the participants, Physical Activity Attitude Scale, International Physical Activity Survey Short Form, Postural Awareness Scale Turkish Version will be used as data collection tools.The Physical Activity Attitude Scale, which was filled out by participants to evaluate their perspectives on physical activity, is a scale consisting of 25 questions with 5 options. It is expressed as "5 = I completely agree, 4 = I mostly agree, 3 = I am undecided, 2 = I slightly agree, 1 = I completely disagree" and a score between 25 and 125 can be obtained. If the total score obtained from the scale is in the range of 25-57, it is considered as low attitude score, if it is in the range of 58-91, it is considered as medium, and if it is in the range of 92-125, it is considered as high attitude score.The International Physical Activity Survey Short Form, which was filled out by participants to determine their physical activity levels, consists of 4 separate sections and a total of 7 questions. The survey asks how many days in the last week and for how long each day heavy physical activity, moderate intensity physical activity and walking were done, and daily sitting time is determined. The total amount of MET spent on these physical activities is calculated. Physical activity levels are classified into 3 different categories: those who are inactive: <600 MET-min/hf, those who are minimally active: >600-3000 MET min/hf, and those who are always active: <3000 MET min/hf.The Turkish Version of the Postural Awareness Scale, which was filled out by the participants to measure their postural awareness level, consists of 11 items, and each item is rated from 1 (not at all applicable to me) to 7 (completely valid for me). Items 1, 2, 3, 4 and 5 of the scale are reverse scored. A minimum of 11 and a maximum of 77 points can be obtained from the scale.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapy and Rehabilitation department or software engineering department is progressing in the 3rd or 4th year undergraduate degree

Exclusion Criteria:

* Having any chronic disease that prevents regular physical activity
* Having a congenital or acquired disease that causes postural disorders and/or having received postural treatment.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physiotherapy and Rehabilitation department or software engineering department is progressing in the 3rd or 4th year undergraduate degree
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-23 (Estimated); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Attitude Scale | 3 months

SECONDARY OUTCOMES:
International Physical Activity Level Short Form Survey | 3 months

OTHER OUTCOMES:
Postural Awareness Scale | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No